CLINICAL TRIAL: NCT01069666
Title: Knowledge Base in the Treatment of Atopic Dermatitis Among Thai Pediatricians
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Pakit Vichyanond, MD, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Other Study IDs: 366/2550(EC3)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Childhood Atopic Dermatitis
Keywords: atopic dermatitis; Thai pediatricians
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine knowledge base in diagnosis, investigation and treatment of pediatric atopic dermatitis among thai pediatricians.

DETAILED DESCRIPTION:
Background: Currently, there is no existing information regarding prescribing practices for the management of childhood atopic dermatitis among pediatricians in Thailand.

Objective: In order to learn about basic knowledge, natural history, evaluation, diagnosis, treatment and prevention for childhood atopic dermatitis in Thailand

Methods: 900 self-administered questionnaires were randomly mailed to pediatricians throughout Thailand, asking about their preferences in the management of childhood atopic dermatitis. One hundred and eighty-five of these 900 questionnaires were returned (a response rate of 20.6%)

ELIGIBILITY:
Inclusion Criteria:

* All pediatricians who're working in thailand including sub-board pediatricians.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 900 self-administered questionnaires were randomly mailed to pediatricians throughout Thailand
Sampling Method: Probability Sample
Dates: Start 2008-07; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Locations (1):
- Facility: Faculty of Medicine Siriraj Hospital, Bangkok, Thailand